CLINICAL TRIAL: NCT06453993
Title: Temporal Variation in Exhaled Volatile Organic Compounds in Response to Therapeutic Intervention in Esophageal Cancer Patients
Brief Title: Temporal Variation in Exhaled Volatile Organic Compounds in Esophageal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRP19015
Record Dates: First submitted 2024-03-11; First posted 2024-06-12 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigate whether exhaled breath can be used to detect and monitor esophageal cancer. (Other): The procedures will include collecting participant's personal information and samples of participant's exhaled breath, urine, and saliva.
  Interventions: Other: Exhaled VOC breath test

INTERVENTIONS:
Other: Exhaled VOC breath test — To determine longitudinal variation in exhaled VOC concentrations during intended curative therapy for EC cancer.

SUMMARY:
The purpose of this study is to investigate whether exhaled breath can be used to detect and monitor esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer ("EG cancer") affects over half a millions people worldwide every year. Early esophageal cancer typically has non-specific symptoms that are often mistaken for benign (non-cancer) conditions. As a result, patients are often referred for further investigations only when they have more prominent symptoms that are typically associated with advanced incurable disease. As a consequence, 7 out of 10 new cases of EG cancer diagnosed are considered to be at an advanced stage, with less than 1 in 3 patients eligible for potentially curative therapy. Better ways of diagnosing esophageal cancer earlier are therefore needed. An ideal test for esophageal cancer would be non-invasive, simple to administer in the community, and cost effective.

The investigators' approach to this clinical challenge is to establish a non-invasive test for the detection of esophageal cancer that is based upon the unique signature of small molecules within exhaled breath. In this study that is being conducted in collaboration with researchers in the United Kingdom (UK), the investigators would like to measure the levels of these small molecules within the breath of patients with esophageal cancer at different times during their treatment: (i) at diagnosis; (ii) after chemoradiotherapy, and; (iii) after surgery. By studying how the small molecules contained within the breath change as a result of esophageal cancer and its treatment, the investigators hope to learn new information that can help develop a new test for this disease.

The investigators will also measure the small molecules within saliva and urine samples collected at the same time as breath in order to study if there are any important differences between these three samples. The investigators will also attempt to measure different bacteria

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90 years
* Newly-diagnosed, treatment naïve patients with esophageal and/or gastroesophageal junctional cancer
* Planning to undergo curative treatment, including neoadjuvant chemoradiotherapy and surgical resection

Exclusion Criteria:

* Pregnant females
* Without malignant esophageal disease
* Malignancy at a secondary site other than the esophagus
* Undergoing palliative treatment for esophageal cancer
* Not receiving neoadjuvant chemoradiotherapy and surgical resection for esophageal cancer
* Inability or unwillingness to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Exhaled breath and urinary VOC concentrations as biomarkers of esophageal cancer | Before commencing treatment for esophageal cancer
  The composition and concentration of volitile organic compounds (VOC) in exhaled breath and urinary samples will be assessed to establish a VOC signature of esophogeal cancer

SECONDARY OUTCOMES:
Changes in VOC concentrations that occur in response to therapeutic intervention | (i) Before commencing treatment for esophageal cancer, (ii) About 4 - 6 weeks after neoadjuvant therapy, (iii) About 3 - 5 days after surgical resection (but before hospital discharge), (iv) At routine follow up (6 - 12 months after surgery)
  VOC concentrations in exhaled breath and urinary samples will be assessed longitudinally to assess how VOC concentrations change in response to therapeutic intervention
Linkage of longitudinal VOC data to predominant upper gastrointestinal bacterial species | (i) Before commencing treatment for esophageal cancer, (ii) About 4 - 6 weeks after neoadjuvant therapy, (iii) About 3 - 5 days after surgical resection (but before hospital discharge), (iv) At routine follow up (6 - 12 months after surgery)
  Bacterial RNA will be extracted from saliva samples to identify bacterial composition. Bacterial composition will then be correlated with breath and urinary VOC levels
Patient acceptability of breath test | Before commencing treatment for esophogeal cancer
  Study subjects will be asked to complete a short survey designed to assess their understanding and opinions regarding breath testing

CONTACTS AND LOCATIONS:
Overall Officials: Donald E Low, MD, Principal Investigator — Virginia Mason Medical Center
Locations (2):
- Virginia Mason Medical Center, Seattle, Washington, United States
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD is not required for analysis. Study ID used to represent study participants.

REFERENCES:
- [Result] Kamal F, Kumar S, Edwards MR, Veselkov K, Belluomo I, Kebadze T, Romano A, Trujillo-Torralbo MB, Shahridan Faiez T, Walton R, Ritchie AI, Wiseman DJ, Laponogov I, Donaldson G, Wedzicha JA, Johnston SL, Singanayagam A, Hanna GB. Virus-induced Volatile Organic Compounds Are Detectable in Exhaled Breath during Pulmonary Infection. Am J Respir Crit Care Med. 2021 Nov 1;204(9):1075-1085. doi: 10.1164/rccm.202103-0660OC. PMID 34319857
- [Result] Antonowicz S, Bodai Z, Wiggins T, Markar SR, Boshier PR, Goh YM, Adam ME, Lu H, Kudo H, Rosini F, Goldin R, Moralli D, Green CM, Peters CJ, Habib N, Gabra H, Fitzgerald RC, Takats Z, Hanna GB. Endogenous aldehyde accumulation generates genotoxicity and exhaled biomarkers in esophageal adenocarcinoma. Nat Commun. 2021 Mar 5;12(1):1454. doi: 10.1038/s41467-021-21800-5. PMID 33674602

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT06453993/Prot_000.pdf
  • Informed Consent Form (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT06453993/ICF_001.pdf